CLINICAL TRIAL: NCT05284149
Title: Study the Impact of Hirsutella Sinensis Nutrient Supplements Has on Improving Muscle Health and Metabolism in Elderly
Acronym: HSN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: Grape King Bio Ltd. (Industry)
Responsible Party: Principal Investigator, Yu-Hsiang Juan, Associate Professor, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 202100881A3
Record Dates: First submitted 2021-12-22; First posted 2022-03-17 (Actual); Last update posted 2022-03-17 (Actual); Status verified 2022-03

CONDITIONS: Sarcopenia; Old Age; Debility; Muscle Loss
MeSH Terms: conditions — Sarcopenia; Frailty; Muscular Atrophy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- H.S. Supplement (Active Comparator): Patients taking Hirsutella Sinensis Nutrient Supplements
  Interventions: Dietary Supplement: Hirsutella Sinensis Nutrient Supplements
- Placebo (Placebo Comparator): Patients taking placebo
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Hirsutella Sinensis Nutrient Supplements — This randomized control study will be conducted in 2 years. We expect to recruit 50 participants with age ≥ 50 years old. Enrolled participants will be recruited into Hirsutella Sinensis nutrient supplement group (50 patients H.S. suppl.) . The medication will be given to the participants by a third party.
  All participants will have two different follow-up periods (6, 12 months). These follow-ups included clinical, laboratory, and imaging studies to analyze muscle health changes after receiving Hirsutella Sinensis nutrient supplement.
  Arms: H.S. Supplement
Dietary Supplement: Placebo — We expect to recruit 50 placebo participants with age ≥ 50 years old. This randomized control study will be conducted in 2 years. The placebo will be given to the participants by a third party.
  All participants will have two different follow-up periods (6, 12 months). These follow-ups included clinical, laboratory, and imaging studies to analyze muscle health changes after receiving placebo.
  Arms: Placebo

SUMMARY:
Sarcopenia has now been officially recognized as a muscle disease related to aging, which may increase the risk of falls and fractures and both heart and respiratory diseases in the elderly. Sarcopenia causes inconvenience in the elderly, affecting their quality of life and often requiring long-term care or even resulting in death. Moreover, the elderly often encountered malnutrition due to inadequate nutrient intake and scarce nutrient diversity. Furthermore, malnutrition is often one of the leading causes of sarcopenia. Therefore, effective nutritional supplementation is essential to improve or prevent muscle loss for the elderly.

Cordyceps sinensis is a well-known valuable traditional Chinese medicine and Hirsutella sinensis was an asexual strain of Cordyceps sinensis. Researchers have found that Hirsutella sinensis can help to increase connection between gastrocnemius muscle fibers and spinal nerve under the amyotrophic lateral sclerosis animal disease model. However, culturing conditions for Hirsutella sinensis are extremely difficult and long, one of the key culturing condition is the temperature, must be maintaining at 16-20℃for 45 days. Fortunately, Grape King Biotech has core technology using liquid fermentation which greatly shortened the cultivation time, thus, providing sufficient and safe products to patients.

The investigators designed a randomized placebo-controlled study first to investigate the relationship and clinical impact Hirsutella Sinensis had on muscle mass and function in the elderly. Second, investigate the metabolic impact Hirsutella Sinensis had on muscle mass.

DETAILED DESCRIPTION:
In 1988, Irwin Rosenberg first proposed the term "Sarcopenia" for sarcopenia, which refers to the amount of muscle loss with age. In 2007, the European Working Group on Sarcopenia in Older People (EWGSOP) reached a consensus of three criteria for aging-related sarcopenia: reduced muscle mass after 65 years of age (60 or 65 years according to the criteria set by each country), weakening of muscle strength (using grip strength), and physiological performance (using walking speed)

Sarcopenia has now been officially recognized as a muscle disease related to aging, which may increase the risk of falls and fractures and both heart and respiratory diseases in the elderly. Sarcopenia causes inconvenience in the elderly, affecting their quality of life and often requiring long-term care or even resulting in death. Moreover, there is now considerable evidence that muscle and bone have common genetic, nutritional, lifestyle, and hormonal determinants. Besides, muscle and bone interact with each other to impact bone strength. A possible mechanism is the dynamic loading arises from muscle contractions and the ground impact during weight-bearing activities. In 2009, the term "sarco-osteopenia" was coined to emphasize that both weak bones and weak muscles may contribute to fractures in the elderly. Therefore, treatments related to increasing muscle mass are essential for the elderly to reduce adverse clinical outcomes such as falls and fractures. At present, the most efficient treatment is adequate nutrient intake.

The elderly often encountered malnutrition due to inadequate nutrient intake and scarce nutrient diversity. While malnutrition is often one of the leading causes of sarcopenia. Therefore, effective nutritional supplementation is essential for the elderly. Efficient nutrient supply will improve the symptoms of sarcopenia patients and improve the quality of life. As Taiwan gradually enters the advanced age society, sarcopenia in the elderly is inevitable. Preventing and treating aging-related muscle loss is becoming a crucial issue that everyone must face. However, there is still a scarcely known nutrient supplement that effectively improves muscle health in the elderly. Moreover, to increase the wiliness of the elderly in taking nutrient supplements, the nutrient supplements must be safe and easily assessable nutrient supplement and do not require a physician prescription. In the Asian population, elderlies incline to Chinese medicine supplements.

Cordyceps sinensis is a well-known valuable traditional Chinese medicine. It is the fungi-insect complex from Clavicipitacease and Cordyceps sinensis (Berk.) Sacc. parasitic on the Heptaidae insects' larvae. Cordyceps sinensis are mainly distributed in the high-mountain areas like Tibet, Sichuan, Qinghai, and Gansu. The traditional Chinese medicine of Cordyceps sinensis have recorded its beneficial effects in kidney and lung, replenishing essence, cough relief and reducing sputum. In the 1990s, a group of female marathon runners led by Mr. Ma Jun-ren, commonly known as Ma family army, trained several world-class middle- and long-distance runner which broke 66 domestic and international records in many competitions. There has been suggestion of his secret performance-enhancing recipe, which includes the combination of Cordyceps, turtle essence and other healthcare products to the athletes' diet. This recipe sets off the Cordyceps market demand once more in China. Enormous Cordyceps were harvested and sold at the same time for research and development. The price of naturally found cordyceps become so scarce that the end-price is almost equivalent to the gold. At the same time period, a total of 22 asexual strains involving 13 genera were isolated from the Cordyceps fruiting bodies collected from different regions. Molecular identification of rDNA ITS region and RAPD molecular markers from the fruiting bodies were detailly compared to finally confirmed that Hirsutella sinensis was an asexual strain of Cordyceps sinensis.

Researchers have found that Hirsutella sinensis has many benefits in anti-inflammatory, anti-liver cancer activity, reduces tetrachloride damage, immune regulation, improves Bleomycin-induced lung fibrosis, aristolochic acid or cisplatin induced Kidney damage… and more. More importantly, study have found that Hirsutella sinensis can help to increase connection between gastrocnemius muscle fibers and spinal nerve under the amyotrophic lateral sclerosis animal disease model. However, culturing conditions for Hirsutella sinensis are extremely difficult and long, one of the key culturing condition is the temperature, must be maintaining at 16-20℃ for 45 days. Fortunately, Grape King Biotech has core technology using liquid fermentation which greatly shortened the cultivation time, thus, providing sufficient and safe products to patients.

The investigators hypothesis that Hirsutella Sinensis may be able to increase both muscle mass and function in the elderly. The investigators believed that improving the muscle mass and function in the elderly may improve the elderly with sarcopenia and prevent the elderly from having sarcopenia. Moreover, it is vital to investigate the metabolic muscle change in the elderly under Hirsutella Sinensis nutrient supplement. This will allow the investigators to further understand the mechanism behind Hirsutella Sinensis had on muscle mass and function.

Specific aims The investigators designed a randomized placebo-controlled study first to investigate the relationship and clinical impact Hirsutella Sinensis had on muscle mass and function in the elderly. Second, investigate the metabolic impact Hirsutella Sinensis had on muscle mass.

2.0 Material and method

2.1.1 Research design This proposal aims to perform a comprehensive analysis of the Hirsutella Sinensis nutrient supplement to improve muscle mass and function. This study comprises an interventional clinical trial that will recruit 100 elderly individuals with either sarcopenia or absence of sarcopenia. All elderly will be receiving clinical, laboratory, and imaging evaluation (in 6, 12 months) to compare the outcome between elderly with and without Hirsutella Sinensis nutrient supplements. This study comprised of comprehensive evaluation of nutrition status, muscle health status and muscle metabolic status for each participant. Furthermore, a detailed metabolomic analysis will be performed on these elderlies to understand the possible mechanism for muscle mass changes and function in the elderly receiving Hirsutella Sinensis nutrient supplements. Figure 1 depict the outline of this study.

2.1 Subjects:

2.1.1 Study duration and subjects number This randomized control study will be conducted in 2 years. The investigators expect to recruit 100 participants with age ≥ 50 years old. Enrolled participants will be randomly divided into Hirsutella Sinensis nutrient supplement (H.S. suppl.) or a placebo group according to a standard randomization procedure (1:1). The medication will be mailed to the participants by a third party.

All participants will have two different follow-up periods (6, 12 months). These follow-ups included clinical, laboratory, and imaging studies to analyze muscle health changes after receiving Hirsutella Sinensis nutrient supplement.

2.1.2 The inclusion criteria As previously described

2.2 Clinical examinations The complete outline of clinical nutrition evaluation, bone fragility evaluation and muscle health evaluation were described in Figure 2.

Figure 2. The outline of clinical assessment

Clinicopathological data:

Clinicopathological data were collected, including age, gender, body height, body weight and waist circumference. Subjects were also asked to list all comorbidities and all current medications. Participants were considered smokers if they currently smoked tobacco or had smoked in the past. Participants were considered alcohol drinkers if they reported consuming alcohol four or more times per week.

Clinical nutrition evaluation:

The nutrition indexes were evaluated using anthropometric method (including the body mass index (BMI)), clinical assessment method (Mini-Nutritional Assessment sheet) and laboratory methods (CBC/DC, lipid profile and albumin).

Muscle health examinations Muscle health status evaluation, including total body composition analysis, handgrip strength (HS) test, and Five-Times-Sit-to-Stand (FTSTS) test. Total body composition analysis may provide us with detailed quantification of fat and muscle of the entire body and different regions of interest. Furthermore, the combination of handgrip strength and Five-Times-Sit-to-Stand tests enables us to understand each participant's muscle function.

Total body composition analysis for muscle mass evaluation:

All the scans were performed using a dual-energy fan-beam X-ray absorptiometry.

Handgrip strength for muscle strength evaluation:

Muscle strength was determined by HS, measured by using a dynamometer.

Five-Times-Sit-to-Stand tests for physical performance evaluation:

The FTSTS test was performed in a quiet room and used a standard chair without armrests. The faster of the 2 trials was used as the FTSTS score.

2.3 Metabolomics examinations The blood sample for metabolomic examination will be taken at the same day as the DXA image study.

B. LC-TOFMS analysis 1a. For global metabolites analysis Liquid chromatographic separation will be achieved on a 100 mm×2.1 mm Acquity 1.7 μm C18 column (Waters Corp; Milford, MA, USA) using a ACQUITY TM Ultra Performance Liquid Chromatography system (Waters, USA).

1b. Mass spectrometry Mass spectrometry will be performed on a Waters Q TOFMS or Agilent Q TOF operated in positive or negative ion mode.

C. Ultra-performance liquid chromatography (UPLC)-based amino acid measurement The plasma samples are collected and stored at -80°C until assayed. The AQC derivatization reagent was obtained from the Waters Corporation (Milford, MA, USA).

2.4 Nutrient supplements Enrolled participants will be randomly divided into Hirsutella Sinensis nutrient supplement (H.S. suppl.) or a placebo group according to a standard randomization procedure (1:1). The medication will be mailed to the participants by a third party. Hirsutella Sinensis and placebo nutrient supplement pills will be identical in appearance. Nutrient supplement pills will be taken for six months.

Composition of Hirsutella Sinensis nutrient supplements: whey protein, modified starch, non-dairy creamer, roux, Hirsutella Sinensis mycelium, maltodextrin, salt, glutamate, flavor enhancers, vegetable oil, lactose, hydrolyzed vegetable protein, onion powder, chicken flavour, locust bean gum, turmeric powder.

Composition of placebo: whey protein, modified starch, non-dairy creamer, roux, maltodextrin, salt, glutamate, flavour enhancers, vegetable oil, lactose, hydrolyzed vegetable protein, onion powder, chicken flavour, locust bean gum, turmeric powder.

Suggested use: 1 sachet (38 g) per day, add 1 sachet of nutrient supplements to 140 mL of hot water, stir well and drink carefully.

Statistical analysis To assess the association of Hirsutella sinensis nutrient supplements had on muscle health and muscle metabolism, Pearson correlation was used for analysis. To analyze the effect of several covariates on muscle health, stepwise logistic regression analysis was applied with adjustments for age, BMI, number of co-morbidities, smoking status, and nutritional status. Logistic regression model and t-test will be applied to analysis the effect of the impact of efficient Hirsutella sinensis nutrient supplements had on improving muscle health.

2.5 Potential difficulties

2.5.1 Concern of DXA safety and participant comfort This study will follow the general DXA safety rules with standard protocols. The participant with DXA contraindication will not be included into this study.

2.5.2 Supports on the particpants' enrollment The elderly population of interest included all those aged 60 years or more who were registered as residents of an administrative neighborhood ("Li") of the North District, Keelung City, Taiwan. In the previous study, the investigators have understand the prevalence of sarcopenia is about 20~40% in the Keelung community. Thus, the recruitment of elderlies with or without sarcopenia will not be a big obstacle in this study.

First year AIMs: Study the effect of Hirsutella sinensis nutrient supplements had on muscle health.

Second year AIMs: Study the metabolomic alternation in muscle after taking Hirsutella sinensis nutrient supplements

3.1 Expected schedule

The First Year:

AIMs: Study the effect of Hirsutella sinensis nutrient supplements had on muscle health

A cross-sectional study on: 1. The relationship between Hirsutella sinensis with muscle mass and function. 2. Compared the improvement of muscle health between participants with and without sarcopenia.

Baseline clinical, laboratory and image data will be collected in 100 participants (Table 1)

The Second Year:

AIMs: Study the metabolomic alternation in muscle after taking Hirsutella sinensis nutrient supplements

A cohort study on the metabolomic change in muscle after receiving Hirsutella sinensis.

One year follow-up clinical and image data will be collected in 100 participants.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for inclusion, each participant must fulfill all of the following criteria:

1. Age >50 years old.
2. Negative pregnancy test for women of childbearing potential.
3. Ability to understand and willingness to be enrolled in our study and sign a written informed consent document

Exclusion Criteria:

Participant who has any of the following criteria will be excluded from the trial:

1. Physical or mental inability.
2. Body mass index (BMI) > 35 kg/m2
3. Participants have acute medical conditions (such as bacterial or viral infection or active cardiopulmonary disease) that may be incapable of having regular image study.
4. Participants are under regular steroid or hyperthyroid medications, which may have great impact on the whole-body metabolism.
5. Participants are under-nutrient, and they need to have regular liquid oral nutrition formulas support.
6. Participants not expecting to comply with follow up.
7. Received barium study within a week
8. Participants allergic or unable ingest Hirsutella Sinensis nutrient supplement

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-02-15 (Actual); Primary Completion 2024-02-15 (Estimated); Study Completion 2024-02-15 (Estimated)

PRIMARY OUTCOMES:
The effect of Hirsutella sinensis nutrient supplements had on muscle health | 1 year
  The change in muscle mass (in grams) as assessed by dual-energy fan-beam X-ray absorptiometry.
Metabolite alternations of Hirsutella Sinensis on muscle health | 1 year
  The changes in major metabolite pathways as assessed (such as amino acids, lipids, in m/z) using the metabolomic liquid chromatography coupled to mass. spectrometry (LC-MS)

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung Memorial Hospital, Keelung Branch, Keelung, Taiwan

IPD SHARING:
Plan to Share IPD: No